CLINICAL TRIAL: NCT03006315
Title: Bio-monitoring of Newly Diagnosed Multiple Myeloma Patients Receiving Induction Chemotherapy Using Mobile Wearable Health Devices
Brief Title: Mobile Health Device Study for Myeloma Patients
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16-1662
Record Dates: First submitted 2016-12-20; First posted 2016-12-30 (Estimated); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Multiple Myeloma; Myeloma
Keywords: multiple myeloma; garmin vivofit
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort A: <65 years: Cohort A will be comprised of participants <65 years old and will accrue a total of 20 patients.
  Interventions: Device: Garmin Vivofit device; Behavioral: Mobile Health quality of life assessements
- Cohort B: >/= 65 years: Cohort B will be comprised of participants >/= 65 years and will accrue a total of 20 patients.
  Interventions: Device: Garmin Vivofit device; Behavioral: Mobile Health quality of life assessements

INTERVENTIONS:
Device: Garmin Vivofit device — Participants will be bio-monitored using the Garmin Vivofit mobile wearable device at baseline (at least 1-7 days prior to treatment initiation) and during induction chemotherapy up to completion of 6 cycles. For those patients continuing with ASCT, patients will be bio-monitored up to 90 days post ASCT.
Behavioral: Mobile Health quality of life assessements

SUMMARY:
Enrolled participants health status will be tracked by using a mobile health-monitoring device while undergoing chemotherapy for multiple myeloma.

DETAILED DESCRIPTION:
Newly diagnosed multiple myeloma participants receiving induction chemotherapy will be continuously bio-monitored at baseline (1-7 days prior to treatment initiation) and during induction chemotherapy up to completion of 6 cycles using the Garmin Vivofit wearable device. For those patients continuing with ASCT, patients will be bio-monitored up to 90 days post ASCT. The study will include a total of 40 newly diagnosed multiple myeloma participants in two cohorts with 20 patients in each cohort (Cohort A and B). Cohort A will be comprised of patients <65 years. Cohort B will be comprised of patients >/= 65 years.

ELIGIBILITY:
Inclusion Criteria

Newly diagnosed Multiple Myeloma meeting International Myeloma Working Group (IMWG) criteria (as below) participants with clinical and histological confirmation of diagnosis planning to receive chemotherapy are eligible:

* Newly diagnosed Multiple Myeloma patients will have evidence of underlying end organ damage and/or myeloma defining event attributed to underlying plasma cell proliferative disorder meeting at least one of the following:
* Hypercalcemia: serum calcium >0.25 mmol/L (> 1 mg/dL) above upper limit of normal or ≥ 2.75 mmol/L (11 mg/dL)
* Anemia: hemoglobin value <10 g/dL or > 2 g/dL below lower limit of normal
* Bone disease: ≥ 1 lytic lesions on skeletal X-ray, CT, or PET-CT. For patients with 1 lytic lesion, bone marrow should demonstrate ≥ 10% clonal plasma cells
* Clonal bone marrow plasma cell percentage ≥ 60%
* Involved/un-involved serum free light chain ratio ≥100 and involved free light chain >100 mg/L
* > 1 focal lesion on magnetic resonance imaging study (lesion must be >5 mm) in size
* All study participants will be required to receive primary chemotherapy treatment at a Memorial Sloan Kettering facility, including regional outpatient sites.
* All study participants will be required to have a smart phone or tablet device compatible with the Garmin Vivofit device.

Exclusion Criteria

* Plasma cell leukemia
* POEMS syndrome
* Amyloidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed Multiple Myeloma participants with clinical and histological confirmation of diagnosis planning to receive chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-11-14 (Actual)

PRIMARY OUTCOMES:
Number of patients continuously wearing the device. | 1 year
  Feasibility of using mobile wearable health device

CONTACTS AND LOCATIONS:
Overall Officials: Neha Korde, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org